CLINICAL TRIAL: NCT01711047
Title: A Study to Investigate the Benefit Of Complex Fractionated Atrial Electrogram (CFAE) Ablation in Addition to Circumferential Pulmonary Vein and Linear Ablations in the Treatment of Persistent Atrial Fibrillation. (BOCA)
Brief Title: Benefit of CFAE Ablation
Acronym: BOCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford University Hospitals NHS Trust (Other)
Collaborators: Royal Bournemouth and Christchurch Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09/H0605/97
Record Dates: First submitted 2012-10-12; First posted 2012-10-22 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Persistent Atrial Fibrillation
Keywords: catheter ablation; atrial fibrillation; pulmonary vein isolation; linear ablation; CFAE ablation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PVI + Linear ablation (Active Comparator): Arm A: patients have PVI and roof and mitral isthmus lines
  Interventions: Procedure: Radiofrequency catheter Ablation
- PVI + linear ablation + CFAE (Active Comparator): Arm B: patients have PVI + roof and mitral isthmus lines and CFAE ablation
  Interventions: Procedure: Radiofrequency catheter ablation

INTERVENTIONS:
Procedure: Radiofrequency catheter Ablation — In this arm, catheter ablation would be performed in the left atrium and would include pulmonary vein isolation and linear ablations (roof and mitral isthmus lines)
  Arms: PVI + Linear ablation
Procedure: Radiofrequency catheter ablation — In this arm, catheter ablation would be performed in the left atrium, including pulmonary vein isolation, linear ablations (roof and mitral isthmus lines) and Complex Fractionated Atrial Electrograms (CFAE) ablation.
  Arms: PVI + linear ablation + CFAE

SUMMARY:
The optimal strategy for catheter ablation of persistent atrial fibrillation is not clearly defined. This study investigates if Complex Fractionated Atrial Electrogram (CFAE) ablation in addition to pulmonary vein isolation and linear ablations improves single procedural success rate over a 12 month follow up period.

ELIGIBILITY:
Inclusion Criteria:

* persistent atrial fibrillation

Exclusion Criteria:

* previous catheter or surgical ablation for atrial fibrillation
* pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-03; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Single procedural success rate (free from AF off anti-arrhythmic drugs) | 12 MONTHS

SECONDARY OUTCOMES:
Multiple procedure success rate | 12 months after last ablation
Complication rate | 30 days of procedure
Percentage of AF termination | Time 0
  This information will be recorded immediately after the procedure.
recurrence of atrial fibrillation or organised atrial tachycardia | 12 months after the last procedure
Ablation time | Time 0
  This information will be recorded immediately after the procedure.
Procedure time | Time 0
  This information will be recorded immediately after the procedure

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Royal Bournemouth Hospital, Bournemouth
  - John Radcliffe Hospital, Oxford

REFERENCES:
- [Derived] Wong KC, Paisey JR, Sopher M, Balasubramaniam R, Jones M, Qureshi N, Hayes CR, Ginks MR, Rajappan K, Bashir Y, Betts TR. No Benefit of Complex Fractionated Atrial Electrogram Ablation in Addition to Circumferential Pulmonary Vein Ablation and Linear Ablation: Benefit of Complex Ablation Study. Circ Arrhythm Electrophysiol. 2015 Dec;8(6):1316-24. doi: 10.1161/CIRCEP.114.002504. Epub 2015 Aug 17. PMID 26283145